CLINICAL TRIAL: NCT06401707
Title: PeRampanel fOr Status ePilEpticus pRophylaxis Post-cardiac Arrest
Acronym: PROSPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-39712
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Heart Arrest; Seizures; Status Epilepticus
Keywords: heart arrest; seizure; status epilepticus; prophylaxis
MeSH Terms: conditions — Heart Arrest; Seizures; Status Epilepticus | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Perampanel (Active Comparator): Perampanel oral load of 24mg upon randomization followed by 8mg oral dose daily for four more days (second dose one day after load and total treatment duration is 5 days)
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): Placebo oral load upon randomization followed by daily placebo oral dose administration for four more days (second dose one day after load and total placebo administration duration is 5 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perampanel — Perampanel is a non-competitive AMPA glutamate receptor antagonist.
  Other Names: Fycompa
  Arms: Perampanel
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Brain injury is the main cause of death and disability for patients surviving cardiac arrest resuscitation and seizures are diagnosed in up to a third of these patients. The investigators are proposing a pilot randomized placebo-controlled clinical trial to evaluate the safety and feasibility of perampanel use for post-cardiac arrest status epilepticus (PCARSE) prevention after cardiac arrest.

DETAILED DESCRIPTION:
More than 500,000 Americans have a cardiac arrest every year and 100,000 survive to hospital admission. Brain injury is the main cause of death and disability for patients surviving cardiac arrest resuscitation and seizures are diagnosed in up to a third of these patients. Seizures with or without muscle jerks, i.e. myoclonic seizures, are the most common seizure type after a cardiac arrest. Despite being common, seizures are usually refractory to treatment (post-cardiac arrest refractory status epilepticus) and the vast majority of patients with this diagnosis die. We are proposing a pilot randomized placebo-controlled clinical trial to evaluate the safety and feasibility of perampanel use for PCARSE prevention after cardiac arrest. Perampanel is a non-competitive AMPA glutamate receptor antagonist approved for adjunctive treatment of partial-onset seizures and primary generalized tonic-clonic seizures, however there are no randomized trials in critically ill cardiac arrest patients at risk for seizures. This medication has been used for the management of refractory status epilepticus, including status epilepticus post-cardiac arrest. We will randomize patients to placebo or perampanel after admission to the intensive care unit. The study's primary outcome will be the incidence of severe adverse events. Secondary efficacy and safety endpoints include incidence of seizures and PCARSE, seizure frequency, time to seizure control, number of anti-seizure medications necessary for seizure control, duration of treatment with anesthetics for seizure control, and time to coma awakening. This study will help determine the safety and feasibility of primary seizure prophylaxis after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Non-traumatic, out-of-hospital cardiac arrest
* Comatose on admission - defined as not following commands
* Return of spontaneous circulation (ROSC) within less than 45 minutes from the time of cardiac arrest (defined as the time of 911 or EMS (emergency medical services) witnessed arrest)
* Admission to the intensive care unit at Zuckerberg San Francisco General Hospital

Exclusion Criteria:

* Acute cerebral hemorrhage or infarction
* Pregnancy
* Prisoner
* Severe kidney function impairment with creatinine clearance inferior to 30 ml/min
* Severe liver impairment with liver function tests five times above the upper limit of normal
* Electrographic or electroclinical seizures diagnosis using American Clinical Neurophysiology criteria confirmed by an epileptologist after cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of perampanel | 7 days
  percentage of participants who are able to complete the 5-day course of perampanel or placebo.
Adverse and Serious Adverse Events | 7 days
  percentage of participants with treatment-related adverse and serious adverse events in perampanel or placebo arms.

SECONDARY OUTCOMES:
Incidence of post-cardiac arrest refractory status epilepticus | 7 days
  percentage of participants with post-cardiac arrest refractory status epilepticus in perampanel or placebo arms.
Incidence of post-cardiac arrest seizures | 7 days
  percentage of participants with post-cardiac arrest seizures in perampanel or placebo arms.
Treatment intensity of post-cardiac arrest refractory status epilepticus | 7 days
  number of anti-seizure medications and anesthetics needed for post-cardiac arrest status epilepticus control in perampanel or placebo arms.
Time to start of post-cardiac arrest refractory status epilepticus | 7 days
  percentage of participants with post-cardiac arrest refractory status epilepticus in perampanel or placebo arms.
Neurological function at 180 days | 180 days
  Distribution of modified Rankin Scale (mRS) score at 180 days in perampanel or placebo arms (mRS range 0 to 6, with higher scores indicating worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Edilberto Amorim, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beretta S, Padovano G, Stabile A, Coppo A, Bogliun G, Avalli L, Ferrarese C. Efficacy and safety of perampanel oral loading in postanoxic super-refractory status epilepticus: A pilot study. Epilepsia. 2018 Oct;59 Suppl 2:243-248. doi: 10.1111/epi.14492. Epub 2018 Aug 29. PMID 30159874
- [Background] Hirsch LJ, Fong MWK, Leitinger M, LaRoche SM, Beniczky S, Abend NS, Lee JW, Wusthoff CJ, Hahn CD, Westover MB, Gerard EE, Herman ST, Haider HA, Osman G, Rodriguez-Ruiz A, Maciel CB, Gilmore EJ, Fernandez A, Rosenthal ES, Claassen J, Husain AM, Yoo JY, So EL, Kaplan PW, Nuwer MR, van Putten M, Sutter R, Drislane FW, Trinka E, Gaspard N. American Clinical Neurophysiology Society's Standardized Critical Care EEG Terminology: 2021 Version. J Clin Neurophysiol. 2021 Jan 1;38(1):1-29. doi: 10.1097/WNP.0000000000000806. No abstract available. PMID 33475321
- See also: Trial Website — https://alab.ucsf.edu/clinical-trials-0